CLINICAL TRIAL: NCT06789380
Title: The (Cost-)Effectiveness of Generalist (GIT-PD) Versus Specialist Treatment (MBT/ST) for Severe Personality Disorders (the P-DAET Study): a Pragmatic Randomized Controlled Non-Inferiority Trial.'
Brief Title: The (Cost-)Effectiveness of Generalist Versus Specialist Treatment for Severe Personality Disorders'
Acronym: P-DAET
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Arkin (Industry)
Collaborators: GGZ de Viersprong (Unknown); Ggz Oost Brabant (Other); Stichting Altrecht GGZ (Unknown); Stichting Dimence Group (Unknown); Tilburg University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P-DAET NL86263.028.24 / P2409
Record Dates: First submitted 2025-01-17; First posted 2025-01-23 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Severe Personality Disorder
Keywords: generalist psychotherapy; specialist psychotherapy; personality disorder; AMPD; schema therapy; mentalisation-based treatment; guideline-informed treatment for personality disorders; level of personality functioning; alternative model of personality disorders; GIT-PD; MBT; ST
MeSH Terms: conditions — Personality Disorders | interventions — Schema Therapy; Mentalization-Based Therapy

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to either group A or B.
  Group A will receive the guideline-infomred treastment for personality disorders (GIT-PD).
  Group B receives either mentalization-based treatment (MBT) or schema therapy (ST), depending on local availbility, treatment history and shared-decision making.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Specialist Treatment for Severe Personality Disorders (Active Comparator): Participants will receive specialist treatment for severe personality disorders. Specifically, the type of treatment will be either mentalization-based treatment (MBT) or schema therapy (ST), depending on local availbility, treatment history and shared-decision making. Both MBT and ST must adhere to the protocol and minimum dosage described in respective effect studies published on MBT or ST.
  Interventions: Behavioral: Schema therapy; Behavioral: Mentalization-based treatment
- Generalist Treatment for Severe Personality Disorders (Experimental): Participants will receive a generalist treatment for severe personality disorders. Specificially, the Guideline-Informed Treatment for Personality Disorders (GIT-PD). Sites can only participate in this study, if they offer a GIT-PD programme of lower dosage than the specialist intervention offered at the same site.
  Interventions: Behavioral: Guideline-informed treatment for personality disorders

INTERVENTIONS:
Behavioral: Schema therapy — Schema therapy (ST) is an evidence-based, fully manualized, specialist form of psychotherapy for personality disorders (Bamelis et al., 2014; Sempértegui et al., 2013; Arntz et al., 2022). Eligible programs must adhere to the minimum standards described in the evidence-based literature. ST is an integrative treatment method, originally rooted in cognitive theory, but with additional influences from Gestalt, psychodynamic, and experiential methods. Schema therapy programs may differ in intensity and duration, even at the same site, but must include a minimum of either 40 sessions and/or a duration of 12 to 24 months. In addition, in order to be eligible, a schema therapy program must be of higher intensity or longer duration than the generalist treatment (GIT-PD) offered at the same site.
  Other Names: Schema-focused therapy; SFT
  Arms: Specialist Treatment for Severe Personality Disorders
Behavioral: Mentalization-based treatment — Mentalization-based treatment (MBT) is an evidence-based, fully manualized, specialist form of psychotherapy for personality disorders (Bateman & Fonagy, 2008; Bateman & Fonagy, 2009; Laurenssen et al., 2018; Juul et al., 2023). MBT is rooted in psychodynamic and attachment theory and aims to alter personality pathology by improving mentalizing and enhancing epistemic trust. Eligible programs must adhere to the minimum standards described in the evidence-based literature. MBT programs may differ in intensity and duration, even at the same site, but must include a minimum of either 40 sessions or a duration of 12 to 24 months. In additon, in order to be eligible, an MBT program must be of higher intensity or longer duration than the generalist treatment (GIT-PD) offered at the same site.
  Arms: Specialist Treatment for Severe Personality Disorders
Behavioral: Guideline-informed treatment for personality disorders — GIT-PD is a non-theoretical and non-methodological approach, based upon principles derived from common factors across evidence-based treatments for PD. GIT-PD has a flexible approach, enabling tailoring treatment to clinical needs of different types of patients. The treatment duration (start-end) is 12- 18 months. The treatment consists of three distinct phases. First, an assessment phase. Second, a modular treatment phase that offers either group or individual interventions. Third, a follow-up phase with limited treatment and focus on relapse prevention. In order to be eligible, GIT-PD should be less intensive than specialist psychotherapies offered in the control arm at the same location (i.e. MBT or ST). GIT-PD will not include evidence-based psychotherapy for personality disorders as described in previous RCTs.
  Arms: Generalist Treatment for Severe Personality Disorders

SUMMARY:
The goal of this clinical trial is to investigate if generalist treatment (GIT-PD) is non-inferior in improving level op personality functioning compared to specialist treatment (MBT/ST) in patients with severe personality disorders. The main questions it aims to answer are:

1. Is generalist treatment (GIT-PD) non-inferior in improving level of personality functioning compared to specialist treatment (MBT/ST) in patients suffering from severe personality disorders (PD)?
2. What patient characteristics predict which patients will benefit more from specialist or generalist treatment?

Participants will be randomized to either specialist or generalist treatment. Interventions included in specialist treatment are Mentalization-Based Treatment (MBT) and Schema Therapy (ST). Generalist treatment will be offererd following the principles of the Guideline-Informed Treatment for Personality Disorders (GIT-PD), a principle-driven treatment framework based upon common factors and allowing personalized treatment according to patients' needs. All participating institutions offer GIT-PD and MBT and/or ST. Before, during and after following this treatment participants will complete measurements at 8 distinct time points.

Participants will be asked to:

* complete a range of instruments at baseline to enable the construction of a personalized advantage index to predict treatment response based on patient characteristics
* complete questionnaires at all 7 post-randomization time points
* undergo a semi-structured interview at 3 time points
* follow treatment for personality disorders (either GIT-PD or MBT/ST)

ELIGIBILITY:
Inclusion Criteria:

* 'severe' or 'extreme' personality disorder (PD) according to the alternative model for PDs

Exclusion Criteria:

* IQ < 75
* legal incapacity
* Any mental state disorder that requires prior treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 358 (Estimated)
Dates: Start 2024-10-21 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Level of Personality Functioning Scale - Brief Form 2.0 (LPFS-BF 2.0) | From enrollment to the follow-up assessment 30 months after the start of treatment.
  The LPFS-BF 2.0 is a self-report questionnaire consisting of 12 items (Weekers et al., 2018). Each item reflects a basic underlying impairment related to the 12 features of personality functioning according to Criterium A of the AMPD such as identity, self-direction, intimacy and relational functioning. The LPFS-BF 2.0 offers a severity index for personality pathology making it suitable for measuring treatment effects. Each item is scored on a scale from 1 (=very false or often false) to 4 (=very true or often true). Therefore, participants achieve a total score between 12 and 48 representing the severity of impairment in personality functioning. Data collection is done digitally via Castor or with pen and paper, based on participants preference. Pen and paper results are copied into Castor by hand by research assistants. Raw data is digitalized and stored on a local drive.
Semi-structured Interview for Personality Functioning (STiP-5.1) | From enrollment to the follow-up assessment 30 months after the start of treatment.
  The STiP-5.1 is a semi-structured clinical interview that provides a multi-item assessment of the severity of personality impairments according to the Level of Personal Functioning Scale (LPFS) of the AMPD included in Section III of DSM-5 (APA, 2013). The interviewer should rate the severity of each facet on a scale ranging between 'little to no impairment' (0) to 'extreme impairment' (4). It takes 45 minutes on average to administer the interview. A total score between 0 and 48 is given to indicate the participants global level of personality functioning . We administer the STiP-5.1 at 3 distinct time points. At the start and end of treatment and after 1 year follow up. All interviews are done by blinded research assistants, and the scores are directly logged in Castor. Interviews will be done either face to face or via video call.

SECONDARY OUTCOMES:
Severity Indices of Personality Problems - Short Form (SIPP-SF) | From enrollment to the follow-up assessment 30 months after the start of treatment.
  The SIPP-SF is a dimensional self-report questionnaire measuring the severity of personality pathology by assessing the core components of adaptive personality functioning. The SIPP-SF is designed in line with the concept of personality disorders as defined in the AMPD. Participants rate the 60 items on a 4-point scale ranging from fully disagree (1) to fully agree (4). Data collection is done digitally via Castor or with pen and paper, based on participants preference. Pen and paper results are copied into Castor by hand by research assistants. Raw data is digitalized and stored on a local drive.
Brief Symptom Inventory (BSI) | From enrollment to the follow-up assessment 30 months after the start of treatment.
  The BSI is a self-report questionnaire investigating symptom severity, consisting of 53 items which can be answered using a scale ranging from 1 (not at all) to 5 (extremely). The total score represents the number of symptoms that participants experienced during the past week. A global severity index and sub scores on all 9 domains are calculated by summing the values on all items and dividing by the number of items/domains. Data collection is done digitally via Castor or with pen and paper, based on participants preference. Pen and paper results are copied into Castor by hand by research assistants. Raw data is digitalized and stored on a local drive.
Columbia Suicide Severity Rating Scale Screen Version (C-SSRS) | From enrollment to the follow-up assessment 30 months after the start of treatment.
  Suicidality is assessed using the C-SSRS. This self-report questionnaire covers 6 items and has been recommended by ICHOM as a standard outcome measurement in personality disorder research, due to its adequate psychometric properties (Prevolnik Rupel et al., 2021). The 6 items are answered with either 'yes' or 'no'. The total number of positive answers indicates suicide risk. Data collection is done digitally via Castor or with pen and paper, based on participants preference. Pen and paper results are copied into Castor by hand by research assistants. Raw data is digitalized and stored on a local drive.
SCID-5-PQ | From enrollment to the follow-up assessment 30 months after the start of treatment.
  The SCID-5-PQ (First et al., 2016) is a self-report measure assessing different criteria for DSM-5 personality disorders according to Section II. Participants are presented with 106 items describing whom they are as a person providing them with a dichotomous 'yes' or 'no' answer scheme. Data collection is done digitally via Castor or with pen and paper, based on participants preference. Pen and paper results are copied into Castor by hand by research assistants. Raw data is digitalized and stored on a local drive.
WHO Disability Assessment Schedule (WHODAS 2.0) | From enrollment to the follow-up assessment 30 months after the start of treatment.
  Social and professional functioning will be measured using the WHODAS 2.0 self-report questionnaire, which includes 12 items. This questionnaire has been recommended by ICHOM for its good reliability, adequate validity and high sensitivity to change (Prevolnik Rupel et al., 2021). Participants answer 12 questions across 6 domains on their daily functioning during the last 30 days. Answers across the 6 domains are weighted and summed to create a total score of disability ranging from 0 to 100. Data collection is done digitally via Castor or with pen and paper, based on participants preference. Pen and paper results are copied into Castor by hand by research assistants. Raw data is digitalized and stored on a local drive.
EQ-5D-5L | From enrollment to the follow-up assessment 30 months after the start of treatment.
  The EQ-5D-5L is a self-report questionnaire that covers 5 items measuring quality of life across 5 domains. Answer options consist of 5 levels ranging from 'no problems' to 'extreme problems'. The level indicates the health state for that domain and can be combined into a 5-digit number indicating the overall quality of life of the participant on that day. Data collection is done digitally via Castor or with pen and paper, based on participants preference. Pen and paper results are copied into Castor by hand by research assistants. Raw data is digitalized and stored on a local drive.
Quality of Life Enjoyment and Satisfaction Questionnaire - Short Form (Q-LES-Q-SF) | From enrollment to the follow-up assessment 30 months after the start of treatment.
  The Q-LES-Q-SF is a self-report questionnaire consisting of 16 items.. Participants rate their satisfaction with different aspects of quality of life on a 5-point scale from "not at all or never" (1) to 'frequently or all the time" (5). The possible scores range from 14 to 70 with higher scores indicating greater satisfaction with life (Stevanovic, 2011). Data collection is done digitally via Castor or with pen and paper, based on participants preference. Pen and paper results are copied into Castor by hand by research assistants. Raw data is digitalized and stored on a local drive.
Treatment Inventory of Costs in Patients with psychiatric disorders (TIC-P for Adults) | From enrollment to the follow-up assessment 30 months after the start of treatment.
  The TIC-P for Adults will be used to assess healthcare consumption and productivity loss during the last 3 months. Through 57 items the costs of different types of care are determined, e.g. for medication use, sessions with therapists, doctor's appointments and more indirect costs like loss of productivity and informal care by the participants network. The first section comprises 8 general questions. The second section includes 22 items regarding healthcare consumption. The last part consists of12 items on informal care and productivity loss. Some items feature multiple follow up questions resulting in the total number of 57 items. Data collection is done digitally via Castor or with pen and paper, based on participants preference. Pen and paper results are copied into Castor by hand by research assistants. Raw data is digitalized and stored on a local drive.

OTHER OUTCOMES:
The Childhood Trauma Questionnaire - Short Form (CTQ-SF) | After enrollment at baseline, pre randomisation.
  The CTQ-SF employs 25 items to assess childhood trauma and distinguish between emotional neglect, physical neglect, emotional abuse, physical abuse and sexual abuse (Bernstein et al., 2003). All statements start with "When I was growing up..." and are answered on a 5-point scale ranging from 1 (never true) to 5 (very often true). Data collection is done digitally via Castor or with pen and paper, based on participants preference. Pen and paper results are copied into Castor by hand by research assistants. Raw data is digitalized and stored on a local drive.
PTSD Checklist for DSM-5 (PCL-5) | After enrollment at basline, pre randomisation.
  The PCL-5 aims to screen for post-traumatic stress disorder using 20 items that correspond to the DSM-5 criteria (Blevins et al., 2015). Likewise, the four subscales correspond to the DSM-5's clusters B through E for PTSD. The 20 items are answered on a 4-point scale ranging from 0 (not at all) to 4 (extremely) resulting in scores ranging between 0 and 80. Data collection is done digitally via Castor or with pen and paper, based on participants preference. Pen and paper results are copied into Castor by hand by research assistants. Raw data is digitalized and stored on a local drive.
Autism Spectrum Quotient | After enrollment at baseline, pre randomisation.
  The 5-item version of the Autism Spectrum Quotient (AQ-5) is a very brief screener, which has been derived from the AQ-10. The AQ-5 measures social communication deficits, corresponding to Criterion A of the ASD-diagnosis. The scale has acceptable internal consistency and convergent validity. Items are rated on a 4 point scale ranging from 'definitely disagree' to 'definitely agree'. Data collection is done digitally via Castor or with pen and paper, based on participants preference. Pen and paper results are copied into Castor by hand by research assistants. Raw data is digitalized and stored on a local drive.
the subscale Motivation to Engage of the Treatment Motivation Scales for forensic outpatient treatment (TMS-F) | After enrollment at baseline, pre randomisation.
  Patient commitment to treatment is measured with a selection of items from the subscale Motivation to Engage of the TMS-F. The four items can be rated on a 7-point Likert scale . Data collection is done digitally via Castor or with pen and paper, based on participants preference. Pen and paper results are copied into Castor by hand by research assistants. Raw data is digitalized and stored on a local drive.
Self-Reflection and Insight Scale | After enrollment at baseline, pre randomisation.
  A modified version of the SRIS is used to assess self- reflection and insight. The SRIS contains 20 5-point Likert scale items ranging from 1 (strongly disagree) to 5 (strongly agree). Data collection is done digitally via Castor or with pen and paper, based on participants preference. Pen and paper results are copied into Castor by hand by research assistants. Raw data is digitalized and stored on a local drive.
Locus of Control Scale (IE) | After enrollment at baseline, pre randomisation.
  Internal locus of control, defined as the extent to which a person experiences an outcome as the result of their own behavior or personal characteristics rather than external circumstance, is assessed by the Locus of Control scale (IE) . The IE contains 10 5-point Likert scale items. Data collection is done digitally via Castor or with pen and paper, based on participants preference. Pen and paper results are copied into Castor by hand by research assistants. Raw data is digitalized and stored on a local drive.
Mental Health Continuum - Short Form (MHC-SF) | After enrollment at baseline, pre randomisation.
  The MHC-SF was developed by Keyes (2008) to measure hedonic and eudaimonic well-being, which can be seen as a separate, but related, dimension to mental "ill-being" (Franken et al., 2018; Keyes, 2007). The questionnaire contains 14 items and three dimensions: emotional well-being (3 items), psychological well-being (6 items) and social well-being (5 items). Data collection is done digitally via Castor or with pen and paper, based on participants preference. Pen and paper results are copied into Castor by hand by research assistants. Raw data is digitalized and stored on a local drive.
Social Problems List from Improving Access to Psychological Therapies (IAPT) | After enrollment at baseline, pre randomisation.
  By using the social problems list, derived from the (IAPT) program social problems (e.g., financial problems, housing problem, and unemployment) are assessed (Clark, 2011). Data collection is done digitally via Castor or with pen and paper, based on participants preference. Pen and paper results are copied into Castor by hand by research assistants. Raw data is digitalized and stored on a local drive.
Multidimensional Scale of Perceived Social Support (MSPSS) | After enrollment at baseline, pre randomisation.
  The MSPSS (O'Toole et al 2012) is assessed to investigate perceived support from three sources: significant others, family, and friends. The MSPSS contains 12 items which can be rated on a 7-point Likert scale ranging from 1 (very strongly disagree) to 7 (very strongly agree). Data collection is done digitally via Castor or with pen and paper, based on participants preference. Pen and paper results are copied into Castor by hand by research assistants. Raw data is digitalized and stored on a local drive.
Stigma of Immutability Scale (Wibbelink, 2022) | After enrollment at baseline, pre randomisation.
  PD has been associated to stigma of immutability (Aviram 2006) and we will use the five items scale as developed by Wibbelink et al (2022), measuring the extent to which participants believe that PD is resistant to treatment. Data collection is done digitally via Castor or with pen and paper, based on participants preference. Pen and paper results are copied into Castor by hand by research assistants. Raw data is digitalized and stored on a local drive.
Dutch Reading Test for Adults (NLV) | After enrollment at baseline, pre randomisation.
  Verbal Intelligence will be measured by the Dutch Reading Test for Adults ('NLV'). Psychometric properties have been shown to be satisfactory among various populations (Hermans et al., 2022). Data collection is done digitally via Castor or with pen and paper, based on participants preference. Pen and paper results are copied into Castor by hand by research assistants. Raw data is digitalized and stored on a local drive.
Questionnaire Epistemic Trust (QET) | After enrollment at baseline, pre randomisation.
  By administering the 24-item QET, insight is gained into a person's developmental capacity to accept information as authentic, trustworthy, generalizable and relevant to the self (i.e. epistemic trust; Knapen et al., 2023). The instrument sheds light on four factors, referring to hypervigilance, curiosity/openness, expectation of help and openness to help. Data collection is done digitally via Castor or with pen and paper, based on participants preference. Pen and paper results are copied into Castor by hand by research assistants. Raw data is digitalized and stored on a local drive.
Personality Inventory for DSM-5 - Short Form (PID-5-SF) | After enrollment at baseline, pre randomisation.
  The PID-5-SF is a shortened 100 item version of the original PID-5 (Maples et al., 2015). It measures 25 facets across 5 domains of pathological personality traits, which corresponds to criterium B of the AMPD (American Psychiatric Association, 2022). Data collection is done digitally via Castor or with pen and paper, based on participants preference. Pen and paper results are copied into Castor by hand by research assistants. Raw data is digitalized and stored on a local drive.

CONTACTS AND LOCATIONS:
Overall Officials: Henricus L. Van, Dr., Principal Investigator — Arkin NPI; Joost Hutsebaut, Prof. dr., Study Director — Tilburg University; GGZ de Viersprong; Nathan Bachrach, Dr., Study Chair — Tilburg University; GGZ Oost-Brabant
Locations (5):
- Netherlands (5):
  - GGZ de Viersprong, Halsteren, North Brabant
  - GGZ Oost-Brabant, Helmond, North Brabant
  - Arkin NPI, Amsterdam, North Holland
  - Dimence Group, Almelo, Overijssel
  - Altrecht, Zeist, Utrecht

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Bomhof C, Loffler JP, Brugman S, Lodder P, van den End A, van Dijk MK, van Westen M, van Dam L, Wielaard I, Mensink W, Muskens L, de Moor B, Bachrach N, Van HL, Hutsebaut J. The effectiveness of generalist (GIT-PD) versus specialist treatment (MBT/ST) for severe personality disorders (Personality Disorders Access to Effective Treatment, P-DAET): study protocol of a pragmatic randomised controlled non-inferiority multicentre trial. BMC Psychiatry. 2025 Nov 20;25(1):1107. doi: 10.1186/s12888-025-07550-4. PMID 41267049
- See also: Study website aimed at a broad audience. — https://p-daet.nl/